CLINICAL TRIAL: NCT03109977
Title: First-in-human Imaging With 89Zr-DFO-pertuzumab in Patients With HER2 Positive Malignancies
Brief Title: Imaging With a New Agent That Finds a Cancer Protein Called HER2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-059
Record Dates: First submitted 2017-04-03; First posted 2017-04-12 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: HER2-positive Carcinoma; HER2-positive Primary Malignancy
Keywords: 17-059; Zr-DFO-pertuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zr-DFO-pertuzumab (89Zr-DFO-pertuzumab) PET/CT (Experimental): Zr-DFO-pertuzumab (89Zr-DFO-pertuzumab) PET/CT will be performed in patients with known HER2-positive malignancy. Patients with multifocal disease, as demonstrated on cross-sectional imaging studies, will be preferentially recruited.
  Interventions: Drug: Zr-DFO-pertuzumab PET/CT

INTERVENTIONS:
Drug: Zr-DFO-pertuzumab PET/CT — Zr-DFO-pertuzumab studies will be performed as hybrid PET/CT examinations with known HER2-positive malignancy

SUMMARY:
The purpose of this study is to test if an imaging agent called Zr-DFO-pertuzumab that finds HER2 proteins can be used to take pictures of HER2-positive cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or greater
* Any biopsy proven HER2-positive malignancy. ASCO guidelines will be used to define HER2-positivity for breast cancer. Similar guidelines will be used for other cancer types as appropriate.
* At least one malignant lesion on CT, MR, or FDG PET/CT within 60 days of protocol enrollment
* ECOG performance of 0-2

Exclusion Criteria:

* Life expectancy < 3 months
* Pregnancy or lactation
* Patients who cannot undergo PET/CT scanning because of weight limits. PET/CT scanners may not be able to function with patients over 450 pounds.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events, including vital signs as Assessed by CTCAE v4.0 | 1 year
  Patients will be monitored closely for evidence of adverse events, including vital signs before and after tracer administration. The day after tracer administration, a physician will screen for any side effects requiring treatment. If a severe adverse effect (Common Terminology Criteria for Adverse Events grade 3 or 4) attributable to 89Zr-DFO-pertuzumab occurs in any patient, then further use of 89Zr-DFO-pertuzumab will be suspended and the protocol reviewed with the MSKCC Data Safety Monitoring Committee.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Ulaner, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Slaon-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org